CLINICAL TRIAL: NCT02438683
Title: A Randomized, Double-blind, Double Dummy, Placebo-controlled, Three-way Crossover Study to Assess Cardiac Effects After Single Oral Doses of BI409306 Under Resting and Exercise Conditions in Healthy Male Volunteers
Brief Title: BI 409306 Cardiac Safety Trial in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.28; 2014-005132-34 (EudraCT Number: EudraCT)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Results first posted 2024-09-03 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306

ARMS (3):
- Placebo under resting/exercise conditions (Placebo Comparator): Participants received matching Placebo oral dose with 240 mL of water after a standardized light breakfast on Day 1 and Day 3 under resting/exercise conditions.
  Interventions: Drug: Placebo
- BI 409306 50 mg under resting/exercise conditions (Experimental): Participants received BI 409306 50 mg oral dose with 240 mL of water after a standardized light breakfast on Day 1 and Day 3 under resting/exercise conditions.
  Interventions: Drug: BI 409306
- BI 409306 200 mg under resting/exercise conditions (Experimental): Participants received BI 409306 200 mg oral dose with 240 mL of water after a standardized light breakfast on Day 1 and Day 3 under resting/exercise conditions.
  Interventions: Drug: BI 409306

INTERVENTIONS:
Drug: BI 409306 — high dose, single dose, oral administration
  Arms: BI 409306 200 mg under resting/exercise conditions
Drug: BI 409306 — low dose, single dose, oral administration
  Arms: BI 409306 50 mg under resting/exercise conditions
Drug: Placebo — single dose, oral administration
  Arms: Placebo under resting/exercise conditions

SUMMARY:
This trial will be conducted to further evaluate, in a controlled setting, potential cardiac effects of an anticipated therapeutic and supra-therapeutic dose of BI 409306 under resting and exercise conditions. Since the drug is being developed in part for a disease with an expectedly high number of elderly (AD), the characterization of cardiac safety of BI 409306 is considered to be important for the development of this compound.

This trial will be conducted to further evaluate, in a controlled setting, potential cardiac effects of an anticipated therapeutic and supra-therapeutic dose of BI 409306 under resting and exercise conditions.

Since the drug is being developed in part for a disease with an expectedly high number of elderly (AD), the characterization of cardiac safety of BI 409306 is considered to be important for the development of this compound.

ELIGIBILITY:
Inclusion criteria:

- Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests.

* Age of 18 to 45 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Waist-to-height ratio less than 0.5
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Ready and able to use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the subject information.

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of

  * Systolic blood pressure less than 90 mm Hg or more than140 mmHg
  * Diastolic blood pressure less than 50 mm Hg or more than 90 mmHg
  * Pulse rate less than 45 bpm or more than 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the PK of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Smoker (unless the subject quit smoking for at least 30 days prior to screening)
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Any suicidal ideation of type 2 to 5 on the C-SSRS in the past 12 months (i.e. active suicidal thought, active suicidal thought with method, active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)
* Any lifetime history of suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour).

In addition, the following trial-specific exclusion criteria apply:

* CYP2C19 PM (no treatment allocation)
* History of macular degeneration
* Beard or unwillingness to shave for the trial (to facilitate appropriate measurements during CPX which requires wearing a face mask)
* Physical disability that precludes safe and adequate CPX investigation
* Known latex allergy

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2015-08-12 (Actual); Study Completion 2015-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1289.28.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Actual number of subjects enrolled in fact represents entered / randomized subjects due to the study set up.
Pre-assignment Details: Screening included informed consent, physical examination, vital signs, Holter Electrocardiogram (ECG), ECG, laboratory, demographics, medical history, Columbia Suicide Severity Rating Scale, cardiopulmonary exercise, concomitant therapy, review of inclusion/exclusion criteria. Subjects genotyped as CYP2C19 poor metabolizers were not to be treated.
Groups:
- Placebo /50 mg/ 200 mg of BI 409306: Participants first received matching Placebo 250 mg, after a separation phase of at least 6 days, they then received BI 409306 50 mg with 200 mg matching placebo, again after a separation phase of at least 6 days, they received BI 409306 200 mg with 50 mg matching placebo film-coated tablets. Every treatment is given oral as 2 single doses (with wash-out phase of approximately 48 hours) with 240 mL of water after a standardized light breakfast on Day 1 and Day 3.
- Placebo /200 mg/ 50 mg of BI 409306: Participants first received matching Placebo 250 mg, after a separation phase of at least 6 days, they then received BI 409306 200 mg with 50 mg matching placebo, again after a separation phase of at least 6 days, they received BI 409306 50 mg with 200 mg matching placebo film-coated tablets. Every treatment is given oral as 2 single doses (with wash-out phase of approximately 48 hours) with 240 mL of water after a standardized light breakfast on Day 1 and Day 3.
- 50 mg / Placebo / 200 mg of BI 409306: Participants first received BI 409306 50 mg with 200 mg matching placebo, after a separation phase of at least 6 days, they then received matching Placebo 250 mg, again after a separation phase of at least 6 days, they received BI 409306 200 mg with 50 mg matching placebo film-coated tablets. Every treatment is given oral as 2 single doses (with wash-out phase of approximately 48 hours) with 240 mL of water after a standardized light breakfast on Day 1 and Day 3.
- 50 mg / 200 mg / Placebo of BI 409306: Participants first received BI 409306 50 mg with 200 mg matching placebo, after a separation phase of at least 6 days, they then received BI 409306 200 mg with 50 mg matching placebo, again after a separation phase of at least 6 days, they received matching Placebo 250 mg film-coated tablets. Every treatment is given oral as 2 single doses (with wash-out phase of approximately 48 hours) with 240 mL of water after a standardized light breakfast on Day 1 and Day 3.
- 200 mg / Placebo / 50 mg of BI 409306: Participants first received BI 409306 200 mg with 50 mg matching placebo, after a separation phase of at least 6 days, they then received matching Placebo 250 mg, again after a separation phase of at least 6 days, they received BI 409306 50 mg with 200 mg matching placebo film-coated tablets. Every treatment is given oral as 2 single doses (with wash-out phase of approximately 48 hours) with 240 mL of water after a standardized light breakfast on Day 1 and Day 3.
- 200 mg / 50 mg / Placebo of BI 409306: Participants first received BI 409306 200 mg with 50 mg matching placebo, after a separation phase of at least 6 days, they then received BI 409306 50 mg with 200 mg matching placebo, again after a separation phase of at least 6 days, they received matching Placebo 250 mg film-coated tablets. Every treatment is given oral as 2 single doses (with wash-out phase of approximately 48 hours) with 240 mL of water after a standardized light breakfast on Day 1 and Day 3.
Period: Overall Study
Arm/Group | Placebo /50 mg/ 200 mg of BI 409306 | Placebo /200 mg/ 50 mg of BI 409306 | 50 mg / Placebo / 200 mg of BI 409306 | 50 mg / 200 mg / Placebo of BI 409306 | 200 mg / Placebo / 50 mg of BI 409306 | 200 mg / 50 mg / Placebo of BI 409306
Started | 4 | 3 | 2 | 3 | 4 | 4
Completed | 3 | 3 | 2 | 3 | 4 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) consisted of all subjects who were documented to have taken at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo /50 mg/ 200 mg of BI 409306 | Placebo /200 mg/ 50 mg of BI 409306 | 50 mg / Placebo / 200 mg of BI 409306 | 50 mg / 200 mg / Placebo of BI 409306 | 200 mg / Placebo / 50 mg of BI 409306 | 200 mg / 50 mg / Placebo of BI 409306 | Total
Number analyzed (Participants) | 4 | 3 | 2 | 3 | 4 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.8 (10.9) | 36.0 (9.2) | 31.0 (5.7) | 28.0 (3.0) | 30.3 (8.2) | 37.8 (9.5) | 32.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 3 | 2 | 3 | 4 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 2 | 3 | 4 | 4 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 4 | 3 | 2 | 3 | 3 | 4 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Slope of the Placebo-corrected Change From Baseline of Heart Rate at Rest and Plasma Concentration Between 0 to 10 Hours
Description: Slope of the placebo-corrected change from baseline in resting heart rate (ΔΔHR) vs. plasma concentration of BI 409306, as assessed from 0 to 10 hours (h) after intake of trial medication. The predicted mean value (90% CI) of ΔΔHR at geometric Mean of Cmax of the corresponding dose group is presented in the measured values table. Primary analysis excluded measurement with missing values. Patients with available data were included.
Time Frame: Baseline and up to 10 hours
Population: The pharmacokinetics electrocardiogram set (PKECGS) included all subjects from the electrocardiogram (ECG) set (all subjects in the treated set who had at least 1 baseline and 1 post-baseline assessment in 1 treatment period for at least 1 ECG interval endpoint) who provided at least 1 valid drug plasma concentration and a corresponding ECG or oxygen variable in any period. Patients in the treatment groups are not mutually exclusive.
Measure: Geometric Mean (90% Confidence Interval); unit: beats/min
Groups:
- BI 409306 50 mg Under Resting Conditions: Participants received BI 409306 50 mg oral dose with 240 mL of water after a standardized light breakfast on Day 1 and Day 3 under resting conditions.
- BI 409306 200 mg Under Resting Conditions: Participants received BI 409306 200 mg oral dose with 240 mL of water after a standardized light breakfast on Day 1 and Day 3 under resting conditions.
Arm/Group | BI 409306 50 mg Under Resting Conditions | BI 409306 200 mg Under Resting Conditions
Number analyzed (Participants) | 16 | 16
beats/min | 0.80 [-0.76 to 2.36] | 5.46 [2.44 to 8.49]
Statistical Analysis 1: Comparison: BI 409306 50 mg Under Resting Conditions vs BI 409306 200 mg Under Resting Conditions; The regression model with response variable placebo-corrected HR change from baseline (ddHR) and independent variable Plasma concentration includes a fixed slope effect as well as random intercept and slope estimates for each subject. (Primary analysis); Test type: Other; The covariance structure is No diagonal Factor Analytic FA0(2); Slope = 0.0029, 95% CI 2-sided [0.0012 to 0.0046]

2. Primary Outcome: Maximum Difference to Placebo of the Change From Baseline in Heart Rate at Rest Between 0 to 4 Hours, Per 50 mg Dose Group
Description: For 50 mg dose, the maximal difference in the change from baseline in resting HR for BI 409306 treatment compared with placebo treatment, as assessed from 0 to 4 hours after intake of trial medication (change from baseline in heart rate at rest between 0-4 hours at the time when maximum difference to placebo of the change from baseline was reached). The note "Not Calculated" represents that the endpoint was not planned to be analyzed for the particular arm and category as only pairwise comparisons were built, no difference to placebo is build. Maximum difference reached at 1 hour. Predicted mean changes from baseline (90% Cis) are shown in the measured value table.
Time Frame: Baseline and up to 4 hours
Population: The electrocardiogram analysis set (ECGS) consisted of all subjects in the treated set who had at least 1 baseline and 1 post-baseline assessment (measured at rest) in 1 treatment period for at least 1 ECG interval endpoint. The ECGS was used for all ECG analyses except for those assessing the relationship between plasma concentration and ECG variables. Patients in the treatment groups are not mutually exclusive.
Measure: Least Squares Mean (Standard Error); unit: beats/min
Groups:
- Placebo Under Resting Conditions: Participants received matching Placebo oral dose with 240 mL of water after a standardized light breakfast on Day 1 and Day 3 under resting conditions.
Arm/Group | BI 409306 50 mg Under Resting Conditions | Placebo Under Resting Conditions
Number analyzed (Participants) | 17 | 18
beats/min | 4.33 (1.33) | 0.48 (1.28)
Statistical Analysis 1: Comparison: BI 409306 50 mg Under Resting Conditions vs Placebo Under Resting Conditions; The a repeated measures model included 'period baseline', 'subject baseline' (defined as the arithmetic mean of the 2 period baselines), 'treatment', 'baseline*time' interaction, 'treatment*time' interaction and 'time' as fixed effects and subject as random effect (Primary analysis); Test type: Other; For the repeated effect 'time', the covariance structure was chosen to be unstructured; Mean Difference (Net) = 3.85, 90% CI 2-sided [0.73 to 6.97], Standard Error of Mean 1.75 — Mean Difference (Net) is actually the adjusted mean difference calculated as BI 409306 50 mg minus Placebo

3. Primary Outcome: Maximum Difference to Placebo of the Change From Baseline in Heart Rate at Rest Between 0 to 4 Hours, Per 200 mg Dose Group
Description: For 200 mg dose, the maximal difference in the change from baseline in resting HR for BI 409306 treatment compared with placebo treatment, as assessed from 0 to 4 hours after intake of trial medication (change from baseline in heart rate at rest between 0-4 hours at the time when maximum difference to placebo of the change from baseline was reached). The note "Not Calculated" represents that the endpoint was not planned to be analyzed for the particular arm and category as only pairwise comparisons were built, no difference to placebo is build. Maximum difference reached at 1 hour. Predicted mean changes from baseline (90% Cis) are shown in the measured value table.
Time Frame: Baseline and up to 4 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: beats/min
Arm/Group | BI 409306 200 mg Under Resting Conditions | Placebo Under Resting Conditions
Number analyzed (Participants) | 17 | 18
beats/min | 5.85 (1.35) | 0.92 (1.33)
Statistical Analysis 1: Comparison: BI 409306 200 mg Under Resting Conditions vs Placebo Under Resting Conditions; [analysis description as in outcome 2, analysis 1]; Test type: Other; For the repeated effect 'time', the covariance structure was chosen to be unstructured; Mean Difference (Net) = 4.93, 90% CI 2-sided [1.69 to 8.16], Standard Error of Mean 1.90 — Mean Difference (Net) is actually the adjusted mean difference calculated as BI 409306 200 mg minus Placebo

4. Secondary Outcome: Slope of Placebo-corrected Change From Baseline of Time Between Start of the Q Wave and End of the T Wave in an ECG Corrected for Heart Rate Using the Fridericia Correction Formula (QTcF) at Rest and Plasma Concentration Between 0 to 10 Hours
Description: Slope of placebo-corrected change from baseline in resting Fridericia correction formula QTcF vs. plasma concentration of BI 409306, as assessed from 0 to 10 h after intake of trial medication. The predicted mean value (90% CI) of ΔΔQTcF at geometric Mean of Cmax of the corresponding dose group is presented in the measured values table. Patients with available data were included.
Time Frame: Baseline and up to 10 hours
Population: The pharmacokinetics electrocardiogram set (PKECGS) included all subjects from the electrocardiogram set (ECGS) who provided at least 1 valid drug plasma concentration and a corresponding ECG or oxygen variable in any period. Patients in the treatment groups are not mutually exclusive.
Measure: Geometric Mean (90% Confidence Interval); unit: milliseconds (msec)
Arm/Group | BI 409306 50 mg Under Resting Conditions | BI 409306 200 mg Under Resting Conditions
Number analyzed (Participants) | 16 | 16
milliseconds (msec) | 0.37 [-1.45 to 2.19] | 2.09 [-1.54 to 5.71]
Statistical Analysis 1: Comparison: BI 409306 50 mg Under Resting Conditions vs BI 409306 200 mg Under Resting Conditions; The regression model with response variable placebo-corrected QTcF change from baseline (ddQTcF) and independent variable. Plasma concentration includes a fixed slope effect as well as random intercept and slope estimates for each subject (Primary analysis). The covariance structure is No diagonal Factor Analytic FA0(2); Test type: Other; The covariance structure is No diagonal Factor Analytic FA0(2); Slope = 0.0011, 95% CI 2-sided [-0.0009 to 0.0030]

5. Secondary Outcome: Maximum Difference to Placebo of the Change From Baseline of QTcF at Rest to Placebo Between 0 to 4 Hours, Per 50 mg Dose Group
Description: For 50 mg dose, the maximal difference in the change from baseline in resting Fridericia correction formula QTcF for BI 409306 treatment compared with placebo treatment, as assessed from 0 to 4 hours after intake of trial medication (change from baseline in resting QTcF at rest between 0-4 hours at the time when maximum difference to placebo of the change from baseline was reached). The note "Not Calculated" represents that the endpoint was not planned to be analyzed for the particular arm and category as only pairwise comparisons were built, no difference to placebo is build. Maximum difference reached at 20 minutes. The predicted mean changes from baseline (90% Cis) are shown in the measured value table.
Time Frame: Baseline and up to 4 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | BI 409306 50 mg Under Resting Conditions | Placebo Under Resting Conditions
Number analyzed (Participants) | 17 | 18
milliseconds (msec) | 10.76 (1.39) | 6.22 (1.37)
Statistical Analysis 1: Comparison: BI 409306 50 mg Under Resting Conditions vs Placebo Under Resting Conditions; [analysis description as in outcome 2, analysis 1]; Test type: Other; For the repeated effect 'time', the covariance structure was chosen to be unstructured; Mean Difference (Net) = 4.54, 90% CI 2-sided [3.39 to 5.70], Standard Error of Mean 0.65 — Mean Difference (Net) is actually the adjusted mean difference calculated as BI 409306 50 mg minus Placebo

6. Secondary Outcome: Maximum Difference to Placebo of the Change From Baseline of QTcF at Rest to Placebo Between 0 to 4 Hours, Per 200 mg Dose Group
Description: For 200 mg dose, the maximal difference in the change from baseline in resting Fridericia correction formula QTcF for BI 409306 treatment compared with placebo treatment, as assessed from 0 to 4 hours after intake of trial medication (change from baseline in resting QTcF at rest between 0-4 hours at the time when maximum difference to placebo of the change from baseline was reached). The note "Not Calculated" represents that the endpoint was not planned to be analyzed for the particular arm and category as only pairwise comparisons were built, no difference to placebo is build. Maximum difference reached at 20 minutes. The predicted mean changes from baseline (90% Cis) are shown in the measured value table.
Time Frame: Baseline and up to 4 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | BI 409306 200 mg Under Resting Conditions | Placebo Under Resting Conditions
Number analyzed (Participants) | 17 | 18
milliseconds (msec) | 11.01 (1.42) | 6.28 (1.38)
Statistical Analysis 1: Comparison: BI 409306 200 mg Under Resting Conditions vs Placebo Under Resting Conditions; [analysis description as in outcome 2, analysis 1]; Test type: Other; For the repeated effect 'time', the covariance structure was chosen to be unstructured; Mean Difference (Net) = 4.73, 90% CI 2-sided [1.34 to 8.13], Standard Error of Mean 1.99 — Mean Difference (Net) is actually the adjusted mean difference calculated as BI 409306 200 mg minus Placebo

7. Secondary Outcome: Slope of the Placebo-corrected Maximum Heart Rate During Exercise vs. Plasma Concentration of BI 409306
Description: Slope of the placebo-corrected maximum heart rate during exercise vs. plasma concentration of BI 409306. Patients with available data were included. Exercise testing was completed before gMean Cmax was reached for BI 409306 200 mg arm. The predicted mean value (90% CI) at geometric Mean of Cmax of the corresponding dose group is presented in the measured values table.
Time Frame: 20 minutes and 2 hours 20 minutes after drug intake
Population: The pharmacokinetics electrocardiogram set (PKECGS) included all subjects from the ECGS who provided at least 1 valid drug plasma concentration and a corresponding ECG or oxygen variable in any period. Patients in the treatment groups are not mutually exclusive.
Measure: Geometric Mean (90% Confidence Interval); unit: beats/min
Groups:
- BI 409306 50 mg Under Exercise Conditions: Participants received BI 409306 50 mg oral dose with 240 mL of water after a standardized light breakfast on Day 1 and Day 3 under exercise conditions.
Arm/Group | BI 409306 50 mg Under Exercise Conditions
Number analyzed (Participants) | 16
beats/min | 2.97 [0.80 to 5.14]
Statistical Analysis 1: Comparison: BI 409306 50 mg Under Exercise Conditions; The regression model with response variable placebo-corrected max HR (dHR) and independent variable Plasma concentration includes a fixed slope effect as well as random intercept and slope estimates for each subject. (Primary analysis); Test type: Other; The covariance structure is Unstructured; Slope = 0.0054, 95% CI 2-sided [0.0032 to 0.0076]

8. Secondary Outcome: Slope of the Placebo Corrected Change From Maximum Heart Rate 1 and 5 Minutes After End of Exercise and Plasma Concentration
Description: Slope of the placebo-corrected difference between maximum heart rate (HR) during exercise and recovery HR at 1 and 5 minutes (min) after the end of exercise vs. plasma concentration of BI 409306. The note "Not Calculated" represents that the plasma concentrations 1 min after the end of exercise did not reach gMean Cmax for the perticular arm. Patients with available data were included. The predicted mean value (90% CI) at geometric Mean of Cmax of the corresponding dose group is presented in the measured values table.
Time Frame: 20 minutes and 2 hours 20 minutes after drug intake
Population: The pharmacokinetics electrocardiogram set (PKECGS) included all subjects from the ECGS who provided at least 1 valid drug plasma concentration and a corresponding ECG or oxygen variable in any period. Patients in the treatment groups were not mutually exclusive.
Measure: Geometric Mean (90% Confidence Interval); unit: beats/min
Groups:
- BI 409306 200 mg Under Exercise Conditions: Participants received BI 409306 200 mg oral dose with 240 mL of water after a standardized light breakfast on Day 1 and Day 3 under exercise conditions.
Arm/Group | BI 409306 50 mg Under Exercise Conditions | BI 409306 200 mg Under Exercise Conditions
Number analyzed (Participants) | 16 | 16
beats/min
  Primary analysis - 1 minute after exercise | 2.14 [0.78 to 3.51] | NA [NA to NA] — Not calculated
  Primary analysis - 5 minutes after exercise | 0.58 [-1.07 to 2.23] | -4.79 [-8.21 to -1.37]
Statistical Analysis 1: Comparison: BI 409306 50 mg Under Exercise Conditions vs BI 409306 200 mg Under Exercise Conditions; The regression model with response variable placebo-corrected change from max HR to recovery HR (ddHR) and independent variable Plasma concentration includes a fixed slope effect as well as random intercept estimates for each subject (Primary analysis); Test type: Other; The covariance structure is Unstructured; Slope = -0.0014, 95% CI 2-sided [-0.0036 to 0.0008]
Statistical Analysis 2: Comparison: BI 409306 50 mg Under Exercise Conditions vs BI 409306 200 mg Under Exercise Conditions; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; The covariance structure is Unstructured; Slope = -0.0029, 95% CI 2-sided [-0.0052 to -0.0007]

ADVERSE EVENTS:
Time Frame: From drug administration until end of washout period or end of trial examination, up to 10 days.
Description: The treated set (TS) consisted of all subjects who were documented to have taken at least 1 dose of trial medication.
Groups:
- Placebo Under Exercise Conditions: Participants received matching Placebo oral dose with 240 mL of water after a standardized light breakfast on Day 1 and Day 3 under exercise conditions.
Arm/Group | Placebo Under Resting Conditions | Placebo Under Exercise Conditions | BI 409306 50 mg Under Resting Conditions | BI 409306 50 mg Under Exercise Conditions | BI 409306 200 mg Under Resting Conditions | BI 409306 200 mg Under Exercise Conditions
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 4/20 | 1/20 | 0/20 | 1/19 | 9/19 | 7/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Under Resting Conditions (N=20) | Placebo Under Exercise Conditions (N=20) | BI 409306 50 mg Under Resting Conditions (N=20) | BI 409306 50 mg Under Exercise Conditions (N=19) | BI 409306 200 mg Under Resting Conditions (N=19) | BI 409306 200 mg Under Exercise Conditions (N=19)
Chromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 3 | 2
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2
Visual brightness (Eye disorders) | 0 | 0 | 0 | 0 | 3 | 1
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes